CLINICAL TRIAL: NCT02115542
Title: Multi Institutional Phase II Trial of Single Agent Regorafenib in Refractory Advanced Biliary Cancers
Brief Title: Single Agent Regorafenib in Refractory Advanced Biliary Cancers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-17651
Record Dates: First submitted 2014-04-11; First posted 2014-04-16 (Estimated); Results first posted 2020-01-13 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-09

CONDITIONS: Cancer of the Bile Duct
Keywords: biliary; liver; Refractory Advanced Biliary Cancers; gallbladder cancer; carcinoma; intra-hepatic biliary system; extra-hepatic biliary system; gall bladder; unresectable; locally advanced; metastatic disease; Bile Duct Diseases; Gallbladder Diseases; regorafenib; stivarga; Bay 73-4506; multikinase inhibitor
MeSH Terms: conditions — Bile Duct Neoplasms; Gallbladder Neoplasms; Carcinoma; Neoplasm Metastasis; Bile Duct Diseases; Gallbladder Diseases | interventions — regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Regorafenib Monotherapy (Experimental): Regorafenib is administered as monotherapy during the study. 160 mg once daily (QD) will be administered for 3 weeks on /1 week off. One cycle is 28 days.
  Interventions: Drug: Regorafenib

INTERVENTIONS:
Drug: Regorafenib — Four 40 mg regorafenib tables should be taken in the morning with approximately 8 fluid ounces (240 mL) of water after a low-fat (<30% fat) breakfast.
  Other Names: Stivarga; BAY73-4506

SUMMARY:
The main purpose of this study is to see if regorafenib can help control or decrease cancer size in patients with cancer of the bile duct. Researchers also want to find out if regorafenib is safe and tolerable.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented carcinoma primary to the intra- or extra-hepatic biliary system or gall bladder with clinical and/or radiologic evidence of unresectable, locally advanced or metastatic disease. Patients with ampullary carcinoma are not eligible.
* Have failed no more than 2 prior lines of systemic chemotherapy for advanced biliary cancer. Patients who received adjuvant chemotherapy and had evidence of disease recurrence within 6 months of completion of the adjuvant treatment are also eligible. If patient received adjuvant treatment and had disease recurrence after 6 months, they will only be eligible after failing one line of systemic chemotherapy used to treat the disease recurrence.
* Eastern Cooperative Oncology Group (ECOG) Performance Status Assessment of 0 or 1
* Measurable and non-measurable disease will be allowed.
* Must not have been treated with any vascular endothelial growth factor (VEGF) inhibitors. Prior 5-Fluorouracil (5-FU) or capecitabine treatment is allowed only if given as a radiosensitizer concurrently with radiation therapy at least 12 weeks prior to registration or if given as part of any adjuvant therapy regimen > 6 months prior to study enrollment.
* Life expectancy of at least 12 weeks (3 months)
* For patients who have received prior cryotherapy, radiofrequency ablation, therasphere, ethanol injection, transarterial chemoembolization (TACE) or photodynamic therapy, the following criteria must be met: 28 days have elapsed since that therapy (lesions that have not been treated with local therapy must be present and measureable.
* Able to understand and willing to sign the written informed consent form
* All acute toxic effects of any prior treatment have resolved to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v4.0 Grade 1 or less at the time of signing the Informed Consent Form (ICF).
* Adequate bone marrow and liver function
* Participants can receive 5-FU or capecitabine.
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of study drug.
* Men and women of childbearing potential must agree to use adequate contraception beginning at the signing of the ICF until at least 3 months after the last dose of study drug.
* Able to swallow and retain oral medication

Exclusion Criteria:

* Previous assignment to treatment during this study. Participants permanently withdrawn from study participation will not be allowed to re-enter study.
* Other investigational treatment during or within 21 days before starting study treatment
* Child Pugh B and C
* Uncontrolled hypertension (systolic pressure >140 mm Hg or diastolic pressure > 90 mm Hg [NCI-CTCAE v4.0] on repeated measurement) despite optimal medical management
* Active or clinically significant cardiac disease
* Evidence or history of bleeding diathesis or coagulopathy
* Any hemorrhage or bleeding event ≥ NCI CTCAE Grade 3 within 4 weeks prior to start of study medication
* Participants with thrombotic, embolic, venous, or arterial events, such as cerebrovascular accident (including transient ischemic attacks) deep vein thrombosis or pulmonary embolism within 6 months of informed consent
* Active malignancy except for nonmelanoma skin cancer or in situ cervical cancer. Potential participants surviving a cancer that was curatively treated and without evidence of disease for more than 3 years before the trial are allowed. All cancer treatments must be completed at least 3 years prior to study entry (i.e., signature date of the informed consent form).
* Potential participants with phaeochromocytoma
* Potential participants with severe hepatic impairment (Child-Pugh Class C)
* Known history of human immunodeficiency virus (HIV) infection or current chronic or active hepatitis B or C infection requiring treatment with antiviral therapy.
* Ongoing infection > Grade 2 NCI-CTCAE v4.0
* Symptomatic metastatic brain or meningeal tumors
* Presence of a non-healing wound, non-healing ulcer, or bone fracture
* Renal failure requiring hemo-or peritoneal dialysis
* Patients with seizure disorder requiring medication
* Persistent proteinuria >/= Grade 3 NCI-CTCAE v4.0 (> 3.5 g/24 hours, measured by urine protein:creatinine ratio on a random urine sample)
* Interstitial lung disease with ongoing signs and symptoms at the time of informed consent
* Pleural effusion or ascites that causes respiratory compromise (≥ NCI-CTCAE version 4.0 Grade 2 dyspnea)
* History of organ allograft (including corneal transplant)
* Known or suspected allergy or hypersensitivity to any of the study drugs, study drug classes, or excipients of the formulations given during the course of this trial
* Any malabsorption condition
* Women who are pregnant or breast-feeding
* Any condition which, in the investigator's opinion, makes the potential participant unsuitable for trial participation
* Substance abuse, medical, psychological or social conditions that may interfere with participation in the study or evaluation of the study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2014-06-05 (Actual); Primary Completion 2018-12-10 (Actual); Study Completion 2021-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Kim, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (3):
- United States (3):
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - VCU Massey Cancer Center, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Regorafenib Monotherapy
Started | 39
Completed | 39
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Regorafenib Monotherapy
Number analyzed (Participants) | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 35
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 35
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 39

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) at 6 Months
Description: OS will be defined as the time from starting on trial to date of death due to any cause. The final analysis will be conducted after the follow-time of the last patient exceeds 6 months.
Time Frame: at 6 month follow-up
Population: Patients that were evaluable for efficacy
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Regorafenib Monotherapy
Number analyzed (Participants) | 32
months | 7.9 [0 to 18.7]

2. Secondary Outcome: Disease Control Response (DCR)
Description: DCR defined as Complete Response (CR) + Partial Response (PR)+ Stable Disease (SD). CR: Complete disappearance of all target and non-target lesions (with the exception of lymph nodes mentioned below); No new lesions. PR: Applies only to patients with at least one measurable lesion; Greater than or equal to 30% decrease under baseline of the sum of appropriate diameters of all target measurable lesions; No unequivocal progression of nonmeasurable disease; No new lesions. SD: Does not qualify for CR, PR, Progression or Symptomatic Deterioration.
Time Frame: Post 6 months follow-up, up to 13 months from on treatment per participant
Population: Patients that were evaluable for efficacy
Measure: Number; unit: percentage of patients
Arm/Group | Regorafenib Monotherapy
Number analyzed (Participants) | 32
percentage of patients | 62.5

3. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the duration of time from start of treatment to time of progression or death, whichever comes first.
  Progression - One or more of the following must occur: 20% increase in the sum of appropriate diameters of target measurable lesions over smallest sum observed (over baseline if no decrease during therapy) using the same techniques as baseline, as well as an absolute increase of at least 0.5 cm. Unequivocal progression of non-measurable disease in the opinion of the treating physician (an explanation must be provided). Appearance of any new lesion/site.
Time Frame: Post 6 months follow-up, up to 13 months from on treatment per participant
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Regorafenib Monotherapy
Number analyzed (Participants) | 32
months | 2.8 [1.1 to 4.5]

ADVERSE EVENTS:
Time Frame: From consent to study completion, 3 years 3 months
Arm/Group | Regorafenib Monotherapy
All-Cause Mortality (participants affected / at risk) | 9/39
Serious Adverse Events (participants affected / at risk) | 27/39
Other Adverse Events (participants affected / at risk) | 39/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regorafenib Monotherapy (N=39)
Death NOS (General disorders) | 6 (6)
Gastritis (Gastrointestinal disorders) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1)
Hiccups (Gastrointestinal disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 5 (5)
Fatigue (General disorders) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Thromboembolic event (Vascular disorders) | 1 (1)
Musculoskeletal and connective tissue disorders -Other (Musculoskeletal and connective tissue disorders) | 1 (1) — Callus removed from foot
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Pneumonia
Fever (General disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 2 (2)
Non-cardiac chest pain (General disorders) | 1 (1)
Facial nerve disorder (Nervous system disorders) | 1 (1) — Bells Palsy
Infections and Infestations - Other (Infections and infestations) | 1 (1) — infected blister on foot
Multi-organ failure (General disorders) | 1 (1)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 (1) — Hematochezia
Infections and Infestations - Other (Infections and infestations) | 1 (1) — Cellulitis
Colitis (Gastrointestinal disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Blood bilirubin increased (Infections and infestations) | 2 (2)
Platelet count decreased (Investigations) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Bile duct stenosis (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regorafenib Monotherapy (N=39)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 20 (34)
Mucositis oral (Gastrointestinal disorders) | 17 (27)
Constipation (Gastrointestinal disorders) | 13 (13)
Nausea (Gastrointestinal disorders) | 12 (20)
Vomiting (Gastrointestinal disorders) | 9 (16)
Ascites (Gastrointestinal disorders) | 8 (8)
Diarrhea (Gastrointestinal disorders) | 8 (13)
Dry mouth (Gastrointestinal disorders) | 4 (4)
Bloating (Gastrointestinal disorders) | 2 (2)
Gastritis (Gastrointestinal disorders) | 2 (2)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 2 (3)
Oral dysesthesia (Gastrointestinal disorders) | 2 (2)
Oral pain (Gastrointestinal disorders) | 2 (2)
Colitis (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Gastroparesis (Gastrointestinal disorders) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Periodontal disease (Gastrointestinal disorders) | 1 (1)
Proctitis (Gastrointestinal disorders) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 25 (42)
Fever (General disorders) | 10 (12)
Pain (General disorders) | 8 (12)
Chills (General disorders) | 4 (6)
Non-cardiac chest pain (General disorders) | 4 (4)
Edema limbs (General disorders) | 3 (3)
Flu like symptoms (General disorders) | 3 (3)
General disorders and administration site conditions - other (General disorders) | 1 (1)
Multi-organ faillure (General disorders) | 1 (1)
Alkaline phosphatase increased (Investigations) | 23 (35)
Alkaline aminotransferase increased (Investigations) | 21 (32)
Aspartate aminotransferase increased (Investigations) | 20 (33)
Blood bilirubin increased (Investigations) | 17 (37)
Platelet count decreased (Investigations) | 15 (32)
Lymphocyte count decreased (Investigations) | 14 (31)
Weight loss (Investigations) | 9 (14)
White blood cell decreased (Investigations) | 8 (15)
Neutrophil count decreased (Investigations) | 7 (9)
Creatinine increased (Investigations) | 2 (2)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Investigations - Other (Investigations) | 1 (1)
Lipase increased (Investigations) | 1 (2)
Lymphocyte count increased (Investigations) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 14 (22)
Hypophosphatemia (Metabolism and nutrition disorders) | 13 (22)
Hyponatremia (Metabolism and nutrition disorders) | 12 (12)
Anorexia (Metabolism and nutrition disorders) | 11 (16)
Hypocalcemia (Metabolism and nutrition disorders) | 9 (14)
Dehydration (Metabolism and nutrition disorders) | 7 (9)
Hyperglycemia (Metabolism and nutrition disorders) | 6 (9)
Hyperkalemia (Metabolism and nutrition disorders) | 6 (7)
Hypokalemia (Metabolism and nutrition disorders) | 4 (6)
Hypermagnesemia (Metabolism and nutrition disorders) | 2 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (2)
Hypertension (Vascular disorders) | 22 (48)
Flushing (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 2 (2)
Thromboembolic event (Vascular disorders) | 2 (2)
Hot flashes (Vascular disorders) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 14 (17)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (8)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pamar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 14 (43)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 (11)
Rash acneiform (Skin and subcutaneous tissue disorders) | 4 (7)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Skin and subcutaneous tissue disorders -Other (Skin and subcutaneous tissue disorders) | 2 (4)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 12 (22)
Leukocytosis (Blood and lymphatic system disorders) | 2 (3)
Headache (Nervous system disorders) | 11 (15)
Dizziness (Nervous system disorders) | 4 (5)
Dysgeusia (Nervous system disorders) | 2 (2)
Tremor (Nervous system disorders) | 2 (2)
Facial nerve disorder (Nervous system disorders) | 1 (2)
Radiculitis (Nervous system disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 9 (14)
Sepsis (Infections and infestations) | 3 (3)
Infections and infestations - Other (Infections and infestations) | 2 (2)
Joint infection (Infections and infestations) | 1 (1)
Nail infection (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2)
Confusion (Psychiatric disorders) | 2 (2)
Agitation (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Hallucinations (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1)
Cyctitis noninfective (Renal and urinary disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Renal and urinary disorders - Other (Renal and urinary disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 2 (2)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Reproductive system and breast disorders - Other (Reproductive system and breast disorders) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (2)
Hypothyroidism (Endocrine disorders) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)
Eye disorders - Other (Eye disorders) | 1 (1)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Neoplasms benign, malignant and unspecified -Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-05): https://cdn.clinicaltrials.gov/large-docs/42/NCT02115542/Prot_SAP_000.pdf